CLINICAL TRIAL: NCT01443546
Title: A Randomized Prospective Trial of Dual Trigger Ovulation in Oocyte Donors
Brief Title: Study of Dual Trigger Ovulation in Oocyte Donors
Acronym: DUALTRIGGER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to complete accrual
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1011011394
Record Dates: First submitted 2011-08-23; First posted 2011-09-29 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Infertility
Keywords: oocyte donor; oocyte recipient; ovulation trigger
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- hCG (Active Comparator): standard dose of hCG for ovulation trigger
  Interventions: Drug: HCG
- Lupron Trigger (Active Comparator): Leuprolide acetate 2 mg ovulation trigger
  Interventions: Drug: Lupron Trigger
- Dual Trigger (Experimental): Lupron and hCG combined ovulation trigger
  Interventions: Drug: Dual Trigger

INTERVENTIONS:
Drug: HCG — hCG Trigger
  Arms: hCG
Drug: Lupron Trigger — leuprolide acetate 2 mg SQ
  Arms: Lupron Trigger
Drug: Dual Trigger — a combination of the two drugs in low dosage (leuprolide acetate 2 mg and hCG 1500 IU).
  Arms: Dual Trigger

SUMMARY:
The project is a randomized, controlled, prospective study of oocyte donors comparing the safety and efficacy of triggering ovulation using a combination of two drugs-GnRH agonist and very low dose hCG-versus triggering ovulation with a standard hCG dose alone or a standard GnRH trigger alone.

DETAILED DESCRIPTION:
The study population will consist of young women, age 21 to 34, presenting to our facility with the desire to donate oocytes and who meet FDA and program requirements for donation.

Participants will be randomized to one of the three treatment interventions for triggering ovulation: 1) a standard dose of hCG, 2) leuprolide acetate 2 mg alone, or 3) a combination of the two drugs in low dosage (leuprolide acetate 2 mg and hCG 1500 IU).

Study participants who choose to repeat oocyte donation during the course of the study trial, and who consent to participate in the trial again, will be randomized in a cross-over manner for any subsequent trials.

Following randomization, the clinical care of study subjects will be the same as for non-participant oocyte donors. Participants in all three study arms will undergo standard ovarian stimulation protocol with gonadotropins, standard individualized adjustment of medication dose, standard criteria for administration of the ovulation trigger dose, and standard egg retrieval procedure.

The recipient population will be recruited from women, age 18 to 55, who present to our center wishing to become pregnant using donor oocytes. All prospective participants who meet the Center for Reproductive Medicine (CRM) criteria be recipients of donated eggs will be eligible to participate, should they wish to do so.

If a prospective recipient consents to participate in the study, then she would be matched with either a donor who is not participating in the study (and is receiving one of our standard triggers for ovulation) or a donor who is participating in the study and whose medication to trigger ovulation has been randomized into one of three groups: standard dose hCG, Leuprolide acetate, or a combination of low dose hCG and Leuprolide acetate.

A recipient who chooses to participate in the study will have no additional tests or procedures over the ones that she would normally do in order to receive donated eggs.

ELIGIBILITY:
Inclusion Criteria:

Donors

* Young women, age 21 to 34, presenting to our facility with the desire to donate oocytes and meeting FDA and program requirements for donation.

Recipients

* Women, age 21 to 55, presenting to our facility with the desire to donate oocytes and meeting FDA and program requirements to be recipients of donated eggs.

Exclusion Criteria:

Donors

* Less than 2 ovaries or any other significant ovarian abnormality
* Does not meet current FDA or program requirements for donation.
* A contraindication for the use of gonadotropins (e.g. tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, clinically significant ovarian cysts)
* A contraindication for the use of oral contraceptive pills (h/o thromboembolism, breast cancer, undiagnosed vaginal bleeding)
* Known gene defects, genetic abnormalities or abnormal karyotype
* Contraindication or hypersensitivity to any of the concomitant medication prescribed as part of the treatment regimen in this protocol
* Inability to give informed consent
* Donors who, because of their place of residence or personal situation, would not be able to commit to all required time points including the one extra visit required by study participation.
* The subject has a recent history of/or current epilepsy, thrombophilia, diabetes, cardiovascular, gastro-intestinal, hepatic, renal or pulmonary or auto-immune disease

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical College- Ronald O. Perelman and Claudia Cohen Center for Reproductive Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://ivf.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Human Chorionic Gonadotropin: standard dose of hCG for ovulation trigger
  HCG: hCG Trigger
Period: Overall Study
Arm/Group | Human Chorionic Gonadotropin | Lupron Trigger | Dual Trigger
Started | 9 | 9 | 8
Completed | 9 | 9 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Inconsistency in the Baseline Analysis Population is related to early termination of the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Human Chorionic Gonadotropin | Lupron Trigger | Dual Trigger | Total
Number analyzed (Participants) | 9 | 9 | 8 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 8 | 26
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 8 | 26
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Having Adverse Events
Description: Any donor having a serious complication such as severe hyperstimulation syndrome, ovarian torsion, infection or peritoneal bleeding will be recorded
Time Frame: 1 month
Population: Total of 26 participants were enrolled. Number of subjects enrolled in each arm were below targeted numbers
Measure: Number; unit: participants
Groups:
- hCG Trigger: standard dose of hCG for ovulation trigger
  HCG: hCG Trigger
Arm/Group | hCG Trigger | Dual Trigger | Lupron Trigger
Number analyzed (Participants) | 9 | 8 | 9
participants | 0 | 1 | 0

2. Primary Outcome: Number of Days Post Retrieval Until Subject is Able to Resume Her Usual Activities
Description: Subjects will complete a brief questionnaire on post retrieval day 7. They will state how many days after retrieval they were able to resume their usual activities.
Time Frame: 7 days post retrieval
Population: Data was not completed by study participants so data was not analyzed for comparison
Arm/Group | hCG Trigger | Dual Trigger | Lupron Trigger
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Ovarian Volume
Description: Ovarian volume of both ovaries will be measured by ultrasound on post op day number 7. Measurements will be taken in three different dimensions and volume calculated from those measurements.
Time Frame: 7 days post retrieval
Population: data for ovarian volume was not collected by 3D ultrasound
Arm/Group | hCG Trigger | Lupron Trigger | Dual Trigger
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Mature Oocytes Retrieved
Description: Number of mature oocytes retrieved will assess the efficacy of the intervention
Time Frame: 1 day post ovulation
Population: Data was not completed by study participants so data was not analyzed for comparison
Arm/Group | hCG Trigger | Dual Trigger | Lupron Trigger
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Pregnancies Per Transfer
Description: Pregnancy rate per transfer will be assessed by hCG level on day 14 post retrieval and clinical pregnancy rate will be assessed by ultrasound on day 28 post retrieval. This will additionally assess efficacy of intervention.
Time Frame: 4 weeks post retrieval
Population: Data was not completed by study participants so data was not analyzed for comparison
Arm/Group | hCG Trigger | Lupron Trigger | Dual Trigger
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | hCG Trigger | Dual Trigger | Lupron Trigger
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | hCG Trigger (N=9) | Dual Trigger (N=8) | Lupron Trigger (N=9)
Ovarian hyper stimulation (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hCG Trigger (N=9) | Dual Trigger (N=8) | Lupron Trigger (N=9)
No oocytes retrieved (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) — No oocytes retrieved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No